CLINICAL TRIAL: NCT05123209
Title: Safety and Efficacy Evaluation of IM83 CAR-T Cells for Patients Wirh Advanced Liver Tumors
Brief Title: Safety and Efficacy Evaluation of IM83 CAR-T Cells for Patients With Advanced Liver Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Immunochina Medical Science & Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: YMCART202101
Record Dates: First submitted 2021-09-08; First posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-09

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IM83 CAR-T cells (Experimental)
  Interventions: Biological: IM83 CAR-T cells
- IM83 CAR-T cells +The second-line treatment (Experimental)
  Interventions: Biological: IM83 CAR-T cells; Combination Product: The second-line treatment of liver cancer

INTERVENTIONS:
Biological: IM83 CAR-T cells — 3×10^9 CAR-T cells
Combination Product: The second-line treatment of liver cancer — approved by NMPA
  Arms: IM83 CAR-T cells +The second-line treatment

SUMMARY:
This is a open-label, single center, cohort study to determine the efficacy and safety of IM83 CAR-T cells in patients with advanced Liver Tumors.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old, male or female.
* Patients with advanced hepatocellular carcinoma (HCC) diagnosed by histopathology or cytology, Barcelona stage B-C.
* Progression or intolerance after receiving standardized systematic treatment in the past (at least first-line treatment fails, and PD-1 / PD-L1 drugs can be used).
* Patients in car-t combined treatment group need to have not received the combined drugs before.
* At least one measurable target lesion according to RECIST1.1.
* Tumor cells expressed GPC3 antigen.
* Child Pugh score of liver function ≤ 7.
* ECOG 0-1.
* Estimated survival ≥ 12 weeks;
* Laboratory inspection shall at least meet the following specified indicators:

ANC≥ 1.5 × 10 ^ 9 / L，platelet ≥ 75 × 10 ^ 9 / L ，Hemoglobin ≥ 90 g / L，Serum creatinine ≤ 1.5 ULN，serum bilirubin ≤ 3 ULN，INR≤ 2，AST and ALT)≤ 5.0 ULN，Creatinine clearance rate ≥ 60 ml / min.

* The left ventricular ejection fraction was > 50%.

Exclusion Criteria:

* The researcher has determined that the subject has autoimmune diseases that are not suitable to participate in this study, such as systemic lupus erythematosus, rheumatoid arthritis, ulcerative colitis.
* History of epilepsy or other central nervous system diseases that may affect the test in the judgment of the investigator.
* The washout period of chemotherapy, molecular targeted therapy, immunotherapy, hepatic artery chemoembolization, radiofrequency ablation, radiotherapy for non target lesions or other anti-tumor drugs within 1 week before blood collection is less than 5 half lives.
* Systemic glucocorticoids (local use is allowed) or other immunosuppressants were used within 3 days before apheresis.
* Other incurable malignant tumors in the past 5 years or at the same time, except cervical carcinoma in situ, skin basal cell carcinoma and breast ductal carcinoma in situ.
* The investigator assessed that the subject had poorly controlled pleural effusion, ascites or pericardial effusion.
* Hypertension with poor drug control (systolic blood pressure > 160mmhg and / or diastolic blood pressure > 90mmHg) or cardiovascular and cerebrovascular diseases with clinical significance (such as active) within 6 months before signing the informed consent, such as cerebrovascular accident, myocardial infarction, unstable angina pectoris, or severe arrhythmia, which cannot be controlled by drugs or has potential impact on the study treatment.
* Combined with other serious organic diseases or mental diseases.
* Subjects with HBsAg or HBcAbpositive and peripheral blood HBV DNA titers of >2000 IU/ml (HBsAg positive but HBV DNA titer <2000 IU/ml of peripheral blood and eligible for antiviral treatment according to chronic hepatitis B prevention guideline 2019 Edition). HCV antibody positive and HCV RNA in peripheral blood > 500 IU / ml. Syphilis antibody positive.
* Male subjects who are pregnant or breastfeeding during the screening period, or who plan pregnancy during treatment or within 1 year after the end of treatment, or whose partner plans pregnancy within 1 year after the end of treatment.
* There were active or uncontrollable infections requiring systemic treatment within 1 week before cell apheresis.
* Other researchers believe that it is not suitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-08-24 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and abnormal laboratory test results as assessed by CTCAE V5.0 | Up to 28 days after CAR-T cell infusion

SECONDARY OUTCOMES:
Objective response rate (ORR) | At 28 days, 3 months and 6 months after CAR-T cell infusion
  ORR, defined as the proportion of participants with a complete response or partial response, as determined by the investigator according to RECIST v1.1
Duration of Response (DOR) | Up to 24 weeks after CAR-T cell infusion
  DOR, defined as the time from the first occurrence of a documented objective response to disease progression or death from any cause (whichever occurs first) in Stage 1, as determined by the investigator according to RECIST v1.1
Progression-free survival (PFS) | Up to 24 weeks after CAR-T cell infusion
  PFS, defined as the time from CAR-T cell infusion to the first occurrence of disease progression or death from any cause (whichever occurs first) , as determined by the investigator according to RECIST v1.1
Overall survival (OS) | Up to 24 weeks after CAR-T cell infusion
  OS , defined as the time from CAR-T cell infusion to death from any cause
Plasma levels of α fetoprotein (AFP) cells infusion | At 28 days, 3 months and 6 months after CAR-T cell infusion
Persistence of CAR-T cells (cell counts and cell percentage in peripheral blood) | Up to 24 weeks after CAR-T cell infusion
  The persistence over time of CAR T cells in the peripheral blood as determined by flow cytometry and qPCR.

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA GENERAL HOSPITAL, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No